CLINICAL TRIAL: NCT04000854
Title: Regenerative Treatment of Traumatized Immature Permanent Incisors With Pulp Necrosis: A Prospective Randomized Multicenter Study
Brief Title: Regenerative Treatment of Traumatized Immature Permanent Incisors With Pulp Necrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Eastman Dental Insitute and Hospital (Other); Umeå University (Other)
Responsible Party: Principal Investigator, Georgios Tsilingaridis, Assistant professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Regenerative endo 181116
Record Dates: First submitted 2019-06-24; First posted 2019-06-27 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Regenerative Endodontics in Traumatized Immature Teeth
Keywords: Dental trauma; pulp necrosis; regenerative; endodontics
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Calcium Hydroxide; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium hydroxide (Active Comparator): Root canal dressing with Ca(OH)2 (Calasept)
  Interventions: Drug: Calcium hydroxide (Calacept)
- Chlorhexidine (Active Comparator): Root canal dressing with clorhexidine digluconate 2 % gel
  Interventions: Drug: Calcium hydroxide (Calacept)

INTERVENTIONS:
Drug: Calcium hydroxide (Calacept) — Long-term follow up of pulp regenerative treatment using two different root canal dressings: calcium hydroxide and chlorhexidin digluconate in immature necrotic traumatized incisiors
  Other Names: Clorhexidine digluconate 2 % gel

SUMMARY:
Endodontic management of traumatized immature permanent teeth with pulp necrosis is both a clinical challenge for the dental practitioners and a public health care problem. Even though there are feasible treatment procedures (such as apexification with calcium hydroxide and with Mineral Trioxide Aggregate (MTA), the long-term survival of these teeth is questionable because none of these techniques can provide continuation of root formation and thickening of the dentin walls. As a result, the immature tooth is weak and prone to fracture.

Recently, regenerative endodontic procedures have gained much attention as biologically based treatment alternative to the techniques described above, but the scientific evidence is insufficient. These procedures aim to remove necrotic and damaged tissues and replace those with healthy functioning pulp-dentin complex.

We plan to invite 120 patients to participate in this study. The inclusion criteria will be children between the ages of 7-19 years with traumatized permanent incisors with immature roots and open apices and pulp necrosis. Patients will be recruited from specialist clinics in Stockholm, Västerbotten and Norrbotten. The patients will be treated by specialists in endodontics and pediatric dentistry with regenerative endodontics. During a 5-year follow-up period the most important outcomes are continuous root development and healing of pulp necrosis. Severe traumatic dental injuries leading to severe complication that could result in early tooth loss can have a severe impact on oral health related quality of life. Therefore, regenerative endodontics can have beneficial effect treating these teeth.

ELIGIBILITY:
Inclusion Criteria:

* Traumatized permanent incisors with immature roots and open apices
* pulp necrosis and apical periodontitis (if present)
* No history of received endodontic treatment of the particular tooth
* Pulp space not needed for post or core restoration
* Good compliance of patient and parents
* Ages from 7-19 years and both genders

Exclusion Criteria:

* Traumatized permanent incisors with mature roots with closed apices (< 1 mm)
* Retreatment cases
* Marginal periodontitis
* Root fracture
* Intraoperative factors such as: lack of bleeding from the periapical tissue, exudate in the root canal prior to revascularization
* Allergy to medicaments used for the treatment

Ages: 7 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2023-12-19 (Estimated); Study Completion 2023-12-19 (Estimated)

PRIMARY OUTCOMES:
Apical periodontitis | Change from baseline radiograph at 12 months
  Presence of apical periodontitis on radiographs after intervention using PeriApicalIndex (PAI).(1) Normal periapical structure; (2) small changes in bone struc- ture; (3) changes in bone structure with some mineral loss; (4) periodontitis with well-defined radiolucent area; and (5) severe periodontitis with exacerbating features.
Root development | Change from baseline radiograph at 12 months
  Continous root development after on radiographs after intervention

SECONDARY OUTCOMES:
Clinical symptoms | Change from baseline at 6 months
  Presence of clinical symptoms such as sinus tract, swelling, mobility, sensitivity on palpation and percussion, bacterial load after treatment with different dressing materials, presence of crown discoloration.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Tsilingaridis, pHd, Principal Investigator — Karolinska Institutet
Locations (1):
- Eastmaninstitutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No